CLINICAL TRIAL: NCT03802695
Title: A Phase 1 Dose Escalation and Expansion Study of Orca-Q, an Engineered Donor Graft Derived From Mobilized Peripheral Blood, in Recipients Undergoing Allogeneic Hematopoietic Cell Transplantation for Hematologic Malignancies
Brief Title: A Phase 1 Study of Orca-Q in Recipients Undergoing Allogeneic Transplantation for Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Orca Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OGFT001-001
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Mixed Phenotype Acute Leukemia; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A (Experimental): Recipients with human leukocyte antigen (HLA)-identical related or unrelated or 1-allele mismatched (7/8 alleles) unrelated donor undergoing myeloablative conditioning (MAC); with single- or dual-agent graft-versus-host disease (GVHD) prophylaxis given
  Interventions: Biological: OrcaGraft (Orca-Q)
- Arm B (Experimental): Recipients with haploidentical-related donors undergoing MAC; with single- or dual-agent GVHD prophylaxis given
  Interventions: Biological: OrcaGraft (Orca-Q)
- Arm C (Experimental): Recipients with an HLA-identical related or unrelated donor undergoing MAC; no GVHD prophylaxis given
  Interventions: Biological: OrcaGraft (Orca-Q)
- Arm D (Experimental): Recipients with an HLA-identical related or unrelated donor undergoing non-myeloablative (NMA)/reduced intensity conditioning (RIC); with dual agent GVHD prophylaxis given
  Interventions: Biological: OrcaGraft (Orca-Q)
- Arm E (Experimental): Recipients with 1-allele mismatched (7/8 alleles) unrelated donor undergoing NMA/RIC; with dual-agent GVHD prophylaxis given
  Interventions: Biological: OrcaGraft (Orca-Q)
- Arm F (Experimental): Recipients with haploidentical-related donors undergoing NMA/RIC; with dual-agent GVHD prophylaxis given
  Interventions: Biological: OrcaGraft (Orca-Q)

INTERVENTIONS:
Biological: OrcaGraft (Orca-Q) — engineered donor allograft

SUMMARY:
This study will evaluate the safety, tolerability, and efficacy of engineered donor grafts ("OrcaGraft"/"Orca-Q") in participants undergoing allogeneic hematopoietic cell transplant (alloHCT) transplantation for hematologic malignancies.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age at the time of enrollment:

   1. For MAC with fully matched donor (Arm A with 8/8 donor and Arm C) and NMA/RIC: Age ≥ 12 and ≤ 78 years
   2. For MAC with mismatched donors (Arm A with 7/8 donor and Arm B): Age ≥ 12 and ≤ 65 years
2. Diagnosed acute myeloid, lymphoblastic or mixed phenotype leukemia, or high or very high risk myelodysplastic syndrome (MDS) either in complete remission (CR) or with ≤ 10 percent of blast cells in bone marrow (BM)
3. Indicated for allogeneic hematopoietic stem cell transplant (alloHCT)
4. Matched to a 8/8 or 7/8 related or unrelated donor, or to a related haploidentical donor
5. Estimated glomerular filtration rate (eGFR) > 50 mL/minute (MAC with tacrolimus) or > 30 mL/minute (NMA/RIC or MAC without tacrolimus)
6. Cardiac parameters: Cardiac ejection fraction ≥ 45 percent (MAC) or ≥ 40 percent (NMA/RIC)
7. Diffusing capacity of the lung for carbon monoxide (DLCO) (adjusted for hemoglobin) ≥ 50 percent for MAC or ≥ 40 percent for NMA/RIC
8. Liver function: Total bilirubin < 1.5 times upper limit of normal (ULN) (MAC) or < 3 times ULN (NMA/RIC); alanine transaminase (ALT)/aspartate transaminase (AST) < 3 times ULN (MAC) or < 5 times ULN (NMA/RIC)
9. Participants enrolling on NMA/RIC-alloHCT arms must be deemed unfit for a myeloablative alloHCT per assessment of the principal investigator (PI)

Key Exclusion Criteria:

1. Prior alloHCT
2. Currently receiving corticosteroids or other immunosuppressive therapy except for approved disease-specific therapy for the patient's underlying hematologic malignancy. Topical corticosteroids or oral systemic corticosteroid doses less than or equal to 10 mg/day are allowed
3. Planned donor lymphocyte infusion (DLI)
4. Planned pharmaceutical in vivo or ex vivo T cell depletion, e.g., post-transplant cyclophosphamide (Cy) or alemtuzumab
5. Positive anti-donor HLA antibodies against a mismatched allele in the selected donor
6. Low performance score: For MAC: Karnofsky Performance Score (KPS) < 70 percent, For NMA/RIC: <60 percent
7. High HCT-specific Comorbidity Index (HCT-CI): For MAC > 4, For NMA/RIC >6
8. Uncontrolled bacterial, viral or fungal infections (currently taking antimicrobial therapy and with progression or no clinical improvement) at time of enrollment
9. Seropositive for human immunodeficiency virus (HIV)-1 or -2, human T-lymphotropic virus (HTLV)-1 or -2 or Hepatitis B surface antigen (HbsAg) or anti-Hepatitis C virus (HCV) antibody (Ab)
10. Any uncontrolled autoimmune disease requiring active immunosuppressive treatment
11. Concurrent malignancies or active disease within 1 year, except non-melanoma skin cancers that have been curatively resected. Patients with concurrent indolent hematologic malignancies that do not require active treatment and are under active surveillance only (such as CLL, low-grade lymphomas, smoldering MM, MZL) may be included with the approval of Medical Monitor
12. History of idiopathic or secondary myelofibrosis
13. Women who are pregnant or breastfeeding

Ages: 12 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities through Day +28 (dose escalation) | 28 Days after administration of Orca-Q/OrcaGraft
  Safety and tolerability of Orca-Q (formerly OrcaGraft) in adults undergoing myeloablative allogeneic hematopoietic cell transplantation (MA-alloHCT) will be evaluated by identification of the following dose limiting toxicities: Grade ≥ 3 infusion-related reaction or cytokine release syndrome, Grade ≥ 3 acute GVHD, Any Grade ≥ 3 treatment-related non-hematologic event not clearly related to the underlying malignancy, intercurrent infection, the HCT conditioning regimen, or other pre-existing medical condition
Primary Graft failure through Day +28 (dose expansion) | 28 Days after administration of Orca-Q/OrcaGraft
  Primary graft failure in the dose expansion phase, defined as being alive without recovery of neutrophils during the evaluation period

SECONDARY OUTCOMES:
Neutrophil Engraftment through Day +28 | 28 days after administration of Orca-Q/OrcaGraft
  Neutrophil engraftment defined as an absolute neutrophil count of >/=500/mm3 for 3 consecutive days
Platelet Engraftment through Day +50 | 50 days after administration of Orca-Q/OrcaGraft
  Platelet engraftment is defined as achieving a platelet count > 20,000/mm3 for 3 consecutive days without platelet transfusion in the preceding 7 days, by Day +50
Secondary Graft Failure through Day +100 | 100 days after administration of Orca-Q/OrcaGraft
  Secondary graft failure is defined as neutrophil engraftment followed by subsequent decline in absolute neutrophil counts < 500 cells/μL, unresponsive to growth factor therapy, by Day +100
Acute GVHD through Day +100 | 100 days after administration of Orca-Q/OrcaGraft
  Acute GVHD will be staged and graded per Mount Sinai Acute GvHD International Consortium (MAGIC) Standardization criteria
Chronic GVHD through Day +365 | 365 days after administration of Orca-Q/OrcaGraft
  Chronic GVHD will be diagnosed per 2014 International NIH Chronic GVHD Diagnosis and Staging Consensus Working Group criteria
Incidence of Non-relapse Mortality (NRM) through Day +365 | 365 days after administration of Orca-Q/OrcaGraft
  NRM is defined as death without evidence of disease recurrence
Incidence of Disease Relapse through Day +365 | 365 days after administration of Orca-Q/OrcaGraft
  Recurrence of primary disease for transplant
GVHD-free and Relapse-free Survival (GRFS) through Day +365 | 365 days after administration of Orca-Q/OrcaGraft
  Survival free from GVHD and relapse
Disease-free Survival (DFS) through Day +365 | 365 days after administration of Orca-Q/OrcaGraft
  DFS is the time from date of transplant to death or relapse, whichever comes first.
Overall Survival through Day +365 | 365 days after administration of Orca-Q/OrcaGraft
  OS is defined as the time from the date of transplant to the date of death from any cause or, for surviving patients, to the date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: James S McClellan, MD, PhD, Study Director — Orca Biosystems, Inc.
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - UC Davis, Sacramento, California
  - Stanford Health Care, Stanford, California
  - Emory University, Atlanta, Georgia
  - The University of Kansas Hospital, Kansas City, Kansas
  - Ohio State University, Columbus, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin